CLINICAL TRIAL: NCT00809133
Title: A Phase I Open Label Trial of Continuous Dosing With BIBW 2992 Combined With Paclitaxel and BIBW 2992 Combined With Paclitaxel and Bevacizumab, BIBW 2992 Combined With Carboplatin and BIBW 2992 Combined With Paclitaxel and Carboplatin in Patients With Advanced Solid Tumours
Brief Title: Trial Exploring Afatinib (BIBW 2992) + Paclitaxel (Part A), Afatinib + Paclitaxel + Bevacizumab (Part B), Afatinib + Carboplatin (Part C) and Afatinib+ Paclitaxel +Carboplatin(Part D) in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 1200.12; 2006-005005-55 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Paclitaxel; Carboplatin; Afatinib; Bevacizumab

ARMS (4):
- Part A (Experimental): BIBW2992 + Paclitaxel
  Interventions: Drug: BIBW 2992; Drug: Paclitaxel
- Part B (Experimental): BIBW2992 + Paclitaxel + Bevacizumab
  Interventions: Drug: Paclitaxel; Drug: BIBW2992; Drug: Bevacizumab
- Part C (Experimental): BIBW2992 + Carboplatin
  Interventions: Drug: Carboplatin; Drug: BIBW 2992
- Part D (Experimental): BIBW2992 +Paclitaxel + Carboplatin
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: BIBW 2992

INTERVENTIONS:
Drug: Paclitaxel — Part A and B:80mg/m2 given on Day 1, 8 and 15 of 28 Day cycle.
  Arms: Part B
Drug: Carboplatin — AUC6 given on day 1 of 21 day cycle
  Arms: Part D
Drug: BIBW 2992 — Escalating dose cohorts
  Arms: Part A
Drug: Paclitaxel — Part A and B:80mg/m2 given on Day 1, 8 and 15 of 28 Day cycle.
  Arms: Part A
Drug: BIBW2992 — MTD dose of part A
  Arms: Part B
Drug: Paclitaxel — 175mg/m2 given on Day 1 of 21 Day cycle
  Arms: Part D
Drug: Carboplatin — AUC6 given on day 1 of 21 day cycle
  Arms: Part C
Drug: Bevacizumab — Escalating dose Cohorts - 5mg / kg, 7.5mg / kg and 10mg / kg given Day 1 and Day 15 of a 28 days cycle
  Arms: Part B
Drug: BIBW 2992 — Escalating dose cohorts
  Arms: Part D
Drug: BIBW 2992 — Escalating dose cohorts
  Arms: Part C

SUMMARY:
The main purpose of this study is to assess the optimum dose of the following medications when they are given together:

* BIBW 2992 and paclitaxel (Taxol)
* BIBW 2992 and paclitaxel and bevacizumab (Avastin)
* BIBW 2992 and carboplatin
* BIBW 2992 and paclitaxel and carboplatin The effect of the different drug combinations will also be assessed.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients (patients) with a histologically confirmed diagnosis of malignancy that is now advanced, non-resectable and / or metastatic.
2. Age 18 years old or older.
3. Life expectancy of at least 3 months.
4. Written informed consent that is consistent with ICH-GCP guidelines.
5. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
6. Patients must have recovered from any previous surgery.
7. Adequate organ function including the following:
8. Cardiac left ventricular function with resting ejection fraction greater than or equal to 50%
9. Absolute neutrophil count of greater than or equal to 1,500/microlitres; greater than 2000/microlitres for carboplatin
10. Platelets greater than or equal to 100,000/microlitres
11. Total bilirubin less than or equal to 1.5 mg/dl (<26 micromol /L, SI unit equivalent).
12. AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X institutional upper limit of normal.
13. Creatinine less than or equal to 1.5 mg/dl (less than or equal to 132 micromol per liter, SI unit equivalent).
14. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) for the duration of trial participation. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days of trial enrolment. Breast feeding mothers will be excluded since these agents may be toxic to infants.

Exclusion criteria:

1. Active infectious disease
2. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
3. GI tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease.
4. Significant cardiovascular disease (a history of congestive heart failure requiring therapy, a need for anti-arrhythmic therapy for a ventricular arrhythmia, unstable angina pectoris or myocardial infarction within 6 months prior to trial entry).
5. Patients who require full-dose anticoagulation.
6. Patients not completely recovered from any therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapies to CTC less than or equal to Grade 1. Prior chemotherapy is allowed if completed at least 4 weeks prior to 1st trial treatment (6 weeks for mitomycin C or nitrosoureas) and the patient has recovered from the acute toxicities of that therapy.
7. Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least 8 weeks, no history of cerebral oedema or bleeding in the past 8 weeks and no requirement for steroids or anti-epileptic therapy
8. Persistent Grade 2 or greater neurotoxicity / neuropathy from any cause.
9. Patients on immunosuppressant therapy or with known HIV infection.
10. Treatment with any of the following within 4 weeks of starting trial medication, or during the trial, is not permitted: chemo-, immuno-, radio- (small field palliative radiotherapy is allowed provided this does not represent clear disease progression), biological therapies (including trastuzumab), hormone therapy (excluding LHRH agonists in prostate cancer, or bisphosphonates), or treatment with other investigational drugs.
11. Participation in another clinical trial within the past 4 weeks before start of therapy or concomitantly with this trial.
12. Prior treatment with EGFR targeting therapies or treatment with EGFR- or HER2 inhibiting drugs within the past 4 weeks before start of therapy or concomitantly with this trial.
13. Patients with known or suspected hypersensitivity to any of the trial drugs, their excipients or similar compounds.
14. Patients unable to comply with the protocol.
15. Active alcohol or drug abuse.
16. Patients with known pre-existing interstitial lung disease

    Additional exclusion criteria for patients recruited to cohorts B:
17. Patients with known or suspected hypersensitivity to bevacizumab, its excipients or Chinese hamster ovary cell products or other recombinant human or humanised antibodies.
18. Patients with brain metastases (a brain scan is not required unless the patient shows signs and symptoms of brain metastases and a brain scan is performed to rule out the presence of brain metastases).
19. Patients with intra-abdominal inflammation .
20. Major surgery within 4 weeks of starting treatment or any wound(s) deemed by the investigator to pose a significant risk to the patient in the event of delayed healing.
21. Prior treatment with anthracycline and/or prior radiation to the chest wall ( patients in these categories will only be entered into the study where the investigator deems the benefit to the patient to outweigh the risk).
22. Patients with any of the following conditions: significant hypertension, significant haemoptysis, known brian metastases, thrombotic or haemorrhagic disorders, INR greater than or equal to 1.5 abnormal PTT, therapeutic anti-coagulation, squamous non small cell lung cancer Additional exclusion criteria for patients recruited to cohorts C and D

    * Patients with severe myelosuppression; i.e. absolute neutrophil count less than 2000/microlitres
    * Patients with renal impairment (creatinine clearance less than 60ml per minute by Cockcroft-Gault equation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- United Kingdom (2):
  - 1200.12.4402 Boehringer Ingelheim Investigational Site, London
  - 1200.12.4401 Boehringer Ingelheim Investigational Site, Sutton

REFERENCES:
- [Derived] O'Brien MER, Sarker D, Bhosle J, Thillai K, Yap TA, Uttenreuther-Fischer M, Pemberton K, Jin X, Wiebe S, de Bono J, Spicer J. A phase I study to assess afatinib in combination with carboplatin or with carboplatin plus paclitaxel in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2018 Nov;82(5):757-766. doi: 10.1007/s00280-018-3661-1. Epub 2018 Aug 7. PMID 30088048
- [Derived] Suder A, Ang JE, Kyle F, Harris D, Rudman S, Kristeleit R, Solca F, Uttenreuther-Fischer M, Pemberton K, Pelling K, Schnell D, de Bono J, Spicer J. A phase I study of daily afatinib, an irreversible ErbB family blocker, in combination with weekly paclitaxel in patients with advanced solid tumours. Eur J Cancer. 2015 Nov;51(16):2275-84. doi: 10.1016/j.ejca.2015.07.041. Epub 2015 Aug 18. PMID 26296295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase I open label trial of continuous dosing with BIBW 2992 (Afatinib) combined with Paclitaxel and BIBW 2992 combined with Paclitaxel and Bevacizumab, BIBW 2992 combined with Carboplatin and BIBW 2992 combined with Paclitaxel and Carboplatin in patients with advanced solid tumours.
Pre-assignment Details: This was a dose-escalation trial, using a 3+3 rule based design. Patients were eligible for repeated treatment courses in the absence of clinical disease progression or undue toxicity.
Groups:
- Part A: A20P80 (Afatinib + Paclitaxel): Afatinib (film-coated tablet) 20 mg qd (once daily) was administered orally in combination with Paclitaxel 80 mg/m2 administered as intravenous infusion on Days 1, 8, and 15 of a 28-day cycle.
- Part A: A40P80 (Afatinib + Paclitaxel): Afatinib (film-coated tablet) 40 mg qd (once daily) was administered orally in combination with Paclitaxel 80 mg/m2 administered as intravenous infusion on Days 1, 8, and 15 of a 28-day cycle.
- Part A: A50P80 (Afatinib + Paclitaxel): Afatinib (film-coated tablet) 50 mg qd (once daily) was administered orally in combination with Paclitaxel 80 mg/m2 administered as intravenous infusion on Days 1, 8, and 15 of a 28-day cycle.
- Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab): Afatinib (film-coated tablet) 20 mg qd (once daily) was administered orally in combination with Paclitaxel 80 mg/m2 administered as intravenous infusion on Days 1, 8 and 15 and Bevacizumab 5mg/kg administered as intravenous infusion on Days 1 and 15 of a 28-day cycle.
- Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab): Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in combination with Paclitaxel 80 mg/m2 administered as intravenous infusion on Days 1, 8 and 15 and Bevacizumab 5mg/kg administered as intravenous infusion on Days 1 and 15 of a 28-day cycle.
- Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab): Afatinib (film-coated tablet) 40 mg qd (once daily) was administered orally in combination with Paclitaxel 80 mg/m2 administered as intravenous infusion on Days 1, 8 and 15 and Bevacizumab 5mg/kg administered as intravenous infusion on Days 1 and 15 of a 28-day cycle.
- Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab): Afatinib (film-coated tablet) 20 mg qd (once daily) was administered orally in combination with Paclitaxel 80 mg/m2 administered as intravenous infusion on Days 1, 8 and 15 and Bevacizumab 7.5 mg/kg administered as intravenous infusion on Days 1 and 15 of a 28-day cycle.
- Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab): Afatinib (film-coated tablet) 20 mg qd (once daily) was administered orally in combination with Paclitaxel 80 mg/m2 administered as intravenous infusion on Days 1, 8 and 15 and Bevacizumab 10 mg/kg administered as intravenous infusion on Days 1 and 15 of a 28-day cycle.
- Part C: A20C6 (Afatinib + Carboplatin): Afatinib (film-coated tablet) 20 mg qd (once daily) administered orally in combination with Carboplatin (intravenous infusion) at a dose targeting an AUC (Area Under the Concentration-time curve) of 6 mg/mL min (AUC6) administered on Day 1 of a 21-day cycle.
- Part C: A40C6 (Afatinib + Carboplatin): Afatinib (film-coated tablet) 40 mg qd (once daily) administered orally in combination with Carboplatin (intravenous infusion) at a dose targeting an AUC (Area Under the Concentration-time curve) of 6 mg/mL min (AUC6) administered on Day 1 of a 21-day cycle.
- Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin): Afatinib (film-coated tablet) 20 mg qd (once daily) was administered orally in combination with Carboplatin AUC5 (intravenous infusion) and Paclitaxel 175 mg/m2 (intravenous infusion) which were administered on Day 1 of a 21-day cycle.
- Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin): Afatinib (film-coated tablet) 30 mg qd (once daily) was administered orally in combination with Carboplatin AUC5 (intravenous infusion) and Paclitaxel 175 mg/m2 (intravenous infusion) which were administered on Day 1 of a 21-day cycle.
- Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin): Afatinib (film-coated tablet) 40 mg qd (once daily) was administered orally in combination with Carboplatin AUC5 (intravenous infusion) and Paclitaxel 175 mg/m2 (intravenous infusion) which were administered on Day 1 of a 21-day cycle.
- Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin): Afatinib (film-coated tablet) 20 mg qd (once daily) was administered orally in combination with Carboplatin AUC6 (intravenous infusion) and Paclitaxel 175 mg/m2 (intravenous infusion) which were administered on Day 1 of a 21-day cycle.
Period: Overall Study
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel) | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab) | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin) | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Started | 3 | 7 | 6 | 3 | 5 | 7 | 6 | 8 | 3 | 9 | 6 | 8 | 5 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 6 | 3 | 5 | 7 | 6 | 8 | 3 | 9 | 6 | 8 | 5 | 7
Not completed — Progressive disease | 2 | 5 | 5 | 3 | 4 | 1 | 3 | 3 | 3 | 9 | 5 | 7 | 5 | 4
Not completed — Dose Limiting Toxicity (DLT) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Other adverse event | 1 | 1 | 1 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Consent withdrawn | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other not mentioned above | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel) | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab) | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin) | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin) | Total
Number analyzed (Participants) | 3 | 7 | 6 | 3 | 5 | 7 | 6 | 8 | 3 | 9 | 6 | 8 | 5 | 7 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (12.9) | 53.6 (11.2) | 56.2 (10.5) | 46.0 (11.1) | 59.0 (6.8) | 52.3 (10.4) | 55.0 (20.5) | 56.6 (9.0) | 73.3 (8.3) | 54.4 (14.7) | 52.0 (9.8) | 53.1 (14.2) | 62.4 (11.1) | 64.6 (8.6) | 56.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5 | 3 | 3 | 4 | 5 | 2 | 0 | 4 | 3 | 7 | 1 | 2 | 44
  Male | 1 | 4 | 1 | 0 | 2 | 3 | 1 | 6 | 3 | 5 | 3 | 1 | 4 | 5 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in the First Cycle for the Determination of the Maximum Tolerated Dose (MTD)
Description: Dose limiting toxicity (DLT) was defined as an Adverse Event (AE) or laboratory abnormality considered as related to study treatment.
Time Frame: Cycle 1: 21 days (part C and D) or 28 days (part A and B)
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Number; unit: Participants
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel) | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab) | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin) | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 5 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 5 | 6
Participants | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD of afatinib in selected combination treatments was defined as the highest dose at which no more than 1 out of 6 patients experienced DLTs during the first treatment cycle, i.e. the highest dose with a DLT incidence ≤17%. The MTD was determined separately for Afatinib in combination with Paclitaxel (part A), Afatinib in combination with Paclitaxel and Bevacizumab (part B), Afatinib and Carboplatin (part C), and Afatinib in combination with Paclitaxel and Carboplatin (part D).
  In part C, dose escalation was not continued beyond the dose level A40C6, due to safety and pharmacokinetic considerations and upon mutual agreement between the investigators and the sponsor. Formally, no MTD was determined, however a recommended phase II dose was determined and is presented here.
  0=not maximum tolerated dose, 1=is maximum tolerated dose
  Note, the depicted order of treatment groups is driven by dose level, not by the actual dosing steps.
Time Frame: Cycle 1: 21 days (part C and D) or 28 days (part A and B)
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Number; unit: Units on a scale
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel) | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab) | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin) | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 5 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 5 | 6
Units on a scale | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0

3. Secondary Outcome: Incidence and Intensity of AEs According to the Maximum Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 Grade
Description: Incidence and Intensity of AEs (Adverse Events) graded according to the maximum CTCAE (Common Toxicity Criteria for Adverse Events) grade based on the number of patients with AEs with CTCAE Grade 1-5.
Time Frame: From first drug administration until the end of treatment cycle 1; 21 days (part C and D) or 28 days (part A and B)
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Number; unit: Participants
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel) | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab) | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin) | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 3 | 7 | 6 | 3 | 5 | 7 | 6 | 8 | 3 | 9 | 6 | 8 | 5 | 7
Participants
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 2 | 2 | 3 | 1 | 2 | 1 | 0 | 3 | 0 | 2 | 1 | 0 | 1 | 2
  Grade 3 | 0 | 5 | 3 | 2 | 2 | 3 | 6 | 4 | 1 | 4 | 3 | 6 | 4 | 3
  Grade 4 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 2
  Grade 5 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0

4. Secondary Outcome: Part A: AUCt,ss: Area Under the Concentration-Time Curve of Afatinib in Plasma at Steady State on Day 15
Description: Area under the concentration-time curve of Afatinib in plasma at steady state.
Time Frame: Day 15: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00 and 24:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel)
Number analyzed (Participants) | 3 | 6 | 4
ng*h/mL | 250 (9.63) | 813 (58.4) | 939 (60.0)

5. Secondary Outcome: Part A: Afatinib Cmax,ss on Day 15
Description: Maximum measured concentration of Afatinib in plasma at steady state.
Time Frame: Day 15: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00 and 24:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel)
Number analyzed (Participants) | 3 | 6 | 5
ng/mL | 12.3 (15.5) | 46.0 (61.9) | 63.5 (74.6)

6. Secondary Outcome: Part A: AUC0-24: Area Under the Concentration-Time Curve of Paclitaxel in Plasma Over the Time Interval From Zero Extrapolated to 24 Hours on Day 1 and Day 15
Description: AUC0-24: Area under the concentration-time curve of Paclitaxel in plasma over the time interval from zero extrapolated to 24 hours.
Time Frame: Day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 24:00. Day 15: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 24:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel)
Number analyzed (Participants) | 3 | 6 | 4
ng*h/mL
  Day 1 (N=3, 6, 5) | 1970 (52.2) | 3730 (28.5) | 3260 (30.1)
  Day 15 (N=3, 6, 5) | 3560 (12.6) | 3170 (67.7) | 3950 (51.8)

7. Secondary Outcome: Part A: Paclitaxel Cmax on Day 1 and Day 15
Description: Maximum measured concentration of Paclitaxel in plasma.
Time Frame: as for outcome 6
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel)
Number analyzed (Participants) | 3 | 6 | 5
ng/mL
  Day 1 | 428 (387) | 2090 (37.7) | 1480 (63.1)
  Day 15 | 1880 (42.2) | 1590 (82.2) | 2120 (68.2)

8. Secondary Outcome: Part B: AUCt,ss: Area Under the Concentration-Time Curve of Afatinib in Plasma at Steady State on Day 15
Description: Area under the concentration-time curve of Afatinib in plasma at steady state.
Time Frame: Day 15: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 24:00. There were no analyzable patients for Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab)
Number analyzed (Participants) | 3 | 0 | 4 | 6 | 4
ng*h/mL | 312 (10.3) |  | 829 (56.3) | 336 (60.1) | 142 (132)

9. Secondary Outcome: Part B: Afatinib Cmax,ss on Day 15
Description: Maximum measured concentration of Afatinib in plasma at steady state.
Time Frame: Day 15: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00 and 24:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab)
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6
ng/mL | 20.4 (16.5) | 21.4 (37.8) | 50.4 (52.9) | 22.8 (78.3) | 9.75 (214)

10. Secondary Outcome: Part B: Area Under the Concentration-Time Curve of Paclitaxel in Plasma Over the Time Interval From 0 Extrapolated Upto 24 Hours on Day 1 and Day 15
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab)
Number analyzed (Participants) | 3 | 5 | 4 | 6 | 5
ng*h/mL
  Day 1 | 3760 (53.0) | 3330 (20.8) | 5090 (38.6) | 3810 (32.9) | 3540 (40.3)
  Day 15 | NA (NA) — No descriptive statistics calculated as there were no analyzable subjects. | NA (NA) — No descriptive statistics calculated as there were no analyzable subjects. | 4060 (31.8) | 5290 (45.6) | NA (NA) — No descriptive statistics calculated as there were no analyzable subjects.

11. Secondary Outcome: Part B: Paclitaxel Cmax on Day 1 and Day 15
Description: Maximum measured concentration of Paclitaxel in plasma.
Time Frame: as for outcome 6
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab)
Number analyzed (Participants) | 3 | 6 | 5 | 6 | 5
ng/mL
  Day 1 | 1800 (112) | 1700 (24.2) | 2950 (26.6) | 1920 (38.4) | 1750 (63.1)
  Day 15 | 1490 (19.4) | 1550 (47.4) | 1620 (39.0) | 2730 (48.4) | 2120 (37.3)

12. Secondary Outcome: Part B: Bevacizumab Plasma Concentration
Description: Bevacizumab plasma concentration after infusion of Bevacizumab 5mg/kg after end of 1st and 2nd infusion in Cycle 1.
Time Frame: as for outcome 6
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Median (Inter-Quartile Range); unit: μg/mL
Groups:
- Part B: End of 1st Infusion of Cycle 1; Part B: End of 2nd Infusion of Cycle 1: Dose escalation of Bevacizumab administered as intravenous infusion to 5 mg/kg. Bevacizumab administered on Days 1 and 15 of a 28-day cycle.
Arm/Group | Part B: End of 1st Infusion of Cycle 1 | Part B: End of 2nd Infusion of Cycle 1
Number analyzed (Participants) | 14 | 14
μg/mL | 119 (53.0) [84.2 to 159] | 154 (20.8) [111 to 168]

13. Secondary Outcome: Part C: AUCt,ss: Area Under the Concentration-Time Curve of Afatinib in Plasma at Steady State in Cycle 2
Description: AUCt,ss: Area under the concentration-time curve of Afatinib in plasma at steady state.
Time Frame: Cycle 2, day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00 and 24:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin)
Number analyzed (Participants) | 2 | 3
ng*h/mL | 511 (1.87) | 465 (91.8)

14. Secondary Outcome: Part C: Afatinib Cmax,ss in Cycle 2
Description: Maximum measured concentration of Afatinib in plasma at steady state.
Time Frame: Cycle 2, day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00 and 24:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin)
Number analyzed (Participants) | 2 | 2
ng/mL | 41.7 (28.0) | 44.2 (9.76)

15. Secondary Outcome: Part C: Area Under the Concentration-Time Curve of Carboplatin in Plasma Over the Time Interval From 0 Extrapolated Upto 24 Hours in Cycle 1 and Cycle 2
Description: AUC0-24: Area under the concentration-time curve of Carboplatin in plasma over the time interval from zero extrapolated to 24 hours.
Time Frame: Cycle 1, day 1 and cycle 2, day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 24:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin)
Number analyzed (Participants) | 3 | 9
ng*h/mL
  Cycle 1 (N=3, 9) | 77500 (5.47) | 76800 (16.9)
  Cycle 2 (N=3, 6) | 77600 (7.36) | 75700 (23.6)

16. Secondary Outcome: Part C: Carboplatin Cmax in Cycle 1 and Cycle 2
Description: Maximum measured concentration of Carboplatin in plasma.
Time Frame: Cycle 1, day 1 and cycle 2, day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 24:00
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin)
Number analyzed (Participants) | 3 | 9
ng/mL
  Cycle 1 (N=3, 9) | 15100 (19.3) | 21100 (31.0)
  Cycle 2 (N=3, 6) | 15200 (18.1) | 19600 (26.8)

17. Secondary Outcome: Part D: AUCt,ss: Area Under the Concentration-Time Curve of Afatinib in Plasma at Steady State.
Description: AUCt,ss: Area under the concentration-time curve of Afatinib at steady state.
Time Frame: Cycle 2, day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00 and 24:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 6 | 2 | 2 | 2
ng*h/mL | 326 (60.4) | 454 (61.7) | 506 (14.9) | 119 (0.110)

18. Secondary Outcome: Part D: Afatinib Cmax,ss
Description: Maximum measured concentration of Afatinib in plasma at steady state.
Time Frame: Cycle 2, day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00 and 24:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 7 | 2 | 2 | 2
ng/mL | 18.3 (52.6) | 27.3 (48.4) | 28.1 (4.27) | 6.73 (7.99)

19. Secondary Outcome: Part D: Area Under the Concentration-Time Curve of Paclitaxel in Plasma Over the Time Interval From 0 Extrapolated Upto 23 Hours in Cycle 1 and Cycle 2
Description: AUC0-23: Area under the concentration-time curve of Paclitaxel in plasma over the time interval from zero extrapolated to 23 hours.
Time Frame: Cycle 1, day 1 and cycle 2, day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00 and 23:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 8 | 7 | 5 | 6
ng*h/mL
  Cycle 1 (N=5, 7, 5, 6) | 10400 (21.8) | 13000 (24.9) | 9220 (43.8) | 10200 (19.9)
  Cycle 2 (N=8, 5, 2, 4) | 10700 (32.2) | 14800 (9.78) | 11900 (41.4) | 9270 (53.2)

20. Secondary Outcome: Part D: Paclitaxel Cmax in Cycle 1 and 2
Description: Maximum measured concentration of Paclitaxel in plasma.
Time Frame: Cycle 1, day 1 and cycle 2, day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00 and 24:00
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 8 | 7 | 5 | 6
ng/mL
  Cycle 1 (N=5, 7, 5, 6) | 3710 (23.4) | 4230 (33.7) | 2570 (36.6) | 3020 (29.1)
  Cycle 2 (N=8, 5, 2, 4) | 3620 (50.9) | 4850 (20.7) | 3290 (52.7) | 2590 (92.3)

21. Secondary Outcome: Part D: Area Under the Concentration-Time Curve of Carboplatin in Plasma Over the Time Interval From 0 Extrapolated Upto 24 Hours in Cycle 1 and Cycle 2
Description: as for outcome 15
Time Frame: Cycle 1, day 1 and cycle 2, day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00 and 24:00
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 8 | 7 | 5 | 7
ng*h/mL
  Cycle 1 (N=5, 7, 5, 7) | 69700 (12.4) | 64900 (29.6) | 68700 (17.2) | 81000 (15.3)
  Cycle 2 (N=8, 5, 2, 5) | 65400 (20.9) | 74800 (15.1) | 72100 (27.5) | 90300 (15.7)

22. Secondary Outcome: Part D: Carboplatin Cmax in Cycle 1 and 2
Description: Maximum measured concentration of Carboplatin in plasma.
Time Frame: Cycle 1, day 1 and cycle 2, day 1: -0:05 (hh:mm), 0:00, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00 and 24:00.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 8 | 7 | 5 | 7
ng/mL
  Cycle 1 (N=5, 7, 5, 7) | 16200 (22.9) | 17900 (17.6) | 15600 (28.0) | 18500 (24.3)
  Cycle 2 (N=8, 5, 2, 5) | 17800 (15.8) | 18600 (24.2) | 12800 (0) | 21500 (14.3)

23. Secondary Outcome: Objective Tumour Response (Unconfirmed)
Description: Number of subjects with objective tumour response (unconfirmed).
  Objective Response (OR) was defined as Complete Response (CR) or Partial Response (PR).
Time Frame: From first drug administration until the last trial drug administration, up to 1156 days.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Number; unit: Participants
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel) | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab) | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin) | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 3 | 7 | 6 | 3 | 5 | 7 | 6 | 8 | 3 | 9 | 6 | 8 | 5 | 7
Participants
  Objective response: No | 3 | 3 | 5 | 3 | 4 | 5 | 5 | 7 | 2 | 7 | 4 | 6 | 2 | 6
  Objective response: Yes | 0 | 4 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 2 | 2 | 3 | 1

24. Secondary Outcome: Objective Tumour Response (Confirmed)
Description: Number of subjects with confirmed objective tumour response.
  Objective Response (OR) was defined as Complete Response (CR) or Partial Response (PR). Objective response was to be confirmed by a second tumour assessment at least 4 weeks after the assessment of CR or PR.
Time Frame: From first drug administration until the last trial drug administration, up to 1156 days.
Population: Treated Set: Patients who received at least 1 dose of study treatment were included in the treated set.
Measure: Number; unit: Participants
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel) | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab) | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin) | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Number analyzed (Participants) | 3 | 7 | 6 | 3 | 5 | 7 | 6 | 8 | 3 | 9 | 6 | 8 | 5 | 7
Participants
  Objective response: No | 3 | 3 | 5 | 3 | 5 | 5 | 5 | 8 | 2 | 7 | 4 | 7 | 3 | 7
  Objective response: Yes | 0 | 4 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 2 | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: From first drug administration until 21 days (part C and D) or 28 days (part A and B) after the last trial drug administration in the last treatment cycle, up to 1184 days.
Arm/Group | Part A: A20P80 (Afatinib + Paclitaxel) | Part A: A40P80 (Afatinib + Paclitaxel) | Part A: A50P80 (Afatinib + Paclitaxel) | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab) | Part C: A20C6 (Afatinib + Carboplatin) | Part C: A40C6 (Afatinib + Carboplatin) | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin)
Serious Adverse Events (participants affected / at risk) | 2/3 | 5/7 | 3/6 | 1/3 | 4/5 | 5/7 | 6/6 | 5/8 | 3/3 | 3/9 | 3/6 | 5/8 | 4/5 | 4/7
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 6/6 | 3/3 | 5/5 | 7/7 | 6/6 | 8/8 | 3/3 | 9/9 | 6/6 | 8/8 | 5/5 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: A20P80 (Afatinib + Paclitaxel) (N=3) | Part A: A40P80 (Afatinib + Paclitaxel) (N=7) | Part A: A50P80 (Afatinib + Paclitaxel) (N=6) | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) (N=3) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) (N=5) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) (N=7) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) (N=6) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab) (N=8) | Part C: A20C6 (Afatinib + Carboplatin) (N=3) | Part C: A40C6 (Afatinib + Carboplatin) (N=9) | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) (N=6) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) (N=8) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) (N=5) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin) (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mycobacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: A20P80 (Afatinib + Paclitaxel) (N=3) | Part A: A40P80 (Afatinib + Paclitaxel) (N=7) | Part A: A50P80 (Afatinib + Paclitaxel) (N=6) | Part B: A20P80B5 (Afatinib + Paclitaxel + Bevacizumab) (N=3) | Part B: A30P80B5 (Afatinib + Paclitaxel + Bevacizumab) (N=5) | Part B: A40P80B5 (Afatinib + Paclitaxel + Bevacizumab) (N=7) | Part B: A20P80B7.5 (Afatinib + Paclitaxel + Bevacizumab) (N=6) | Part B: A20P80B10 (Afatinib + Paclitaxel + Bevacizumab) (N=8) | Part C: A20C6 (Afatinib + Carboplatin) (N=3) | Part C: A40C6 (Afatinib + Carboplatin) (N=9) | Part D: A20P175C5 ( Afatinib + Paclitaxel + Carboplatin) (N=6) | Part D: A30P175C5 (Afatinib + Paclitaxel + Carboplatin) (N=8) | Part D: A40P175C5 (Afatinib + Paclitaxel + Carboplatin) (N=5) | Part D: A20P175C6 (Afatinib + Paclitaxel + Carboplatin) (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 2 | 4 | 2 | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 2
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 4 | 5 | 5 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 3 | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Episcleritis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 3 | 0 | 3 | 4 | 3 | 1 | 2 | 3 | 4 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 7 | 6 | 3 | 4 | 6 | 4 | 7 | 1 | 6 | 6 | 6 | 5 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 2 | 2 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 5 | 2 | 4 | 5 | 1 | 6 | 2 | 3 | 3 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 3 | 1 | 3 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 2 | 1 | 2 | 3 | 0 | 4 | 2 | 4 | 1 | 2
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 5 | 5 | 3 | 5 | 6 | 4 | 6 | 3 | 7 | 5 | 5 | 5 | 6
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 5 | 4 | 2 | 2 | 5 | 2 | 5 | 0 | 2 | 2 | 5 | 3 | 3
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 3 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 4 | 1 | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis in device (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 2 | 2 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Omphalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 5 | 0 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 5 | 4 | 0 | 3 | 3 | 3 | 3 | 1 | 4 | 1 | 2 | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 5 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 2 | 2 | 3 | 1 | 1
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brachial plexopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 2 | 3 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 2
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 2 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 4 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 3 | 2 | 3 | 1 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Galactostasis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 1 | 2 | 3 | 1 | 4 | 0 | 2 | 1 | 0 | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 4 | 0 | 2 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 3 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 3 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 3 | 3 | 4 | 3 | 0 | 3 | 1 | 3 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 0 | 3 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 3 | 1 | 1 | 1 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 1 | 3 | 2 | 4 | 4 | 0 | 0 | 3 | 2 | 3 | 5
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0 | 3 | 1 | 1 | 1 | 5 | 3 | 1 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 0 | 4 | 3 | 0 | 1 | 0 | 2 | 2 | 3 | 1 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nail pitting (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 6 | 5 | 3 | 4 | 4 | 3 | 6 | 2 | 2 | 2 | 6 | 5 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.